CLINICAL TRIAL: NCT02339389
Title: Does Maternal Fever During Labor Analgesia Has Any Relationship With Maternal Ventilation?
Acronym: matvent
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Bhavani Shankar Kodali, Interim Chairman, Anesthesiology, Brigham and Women's Hospital
Other Study IDs: 2014P00152
Record Dates: First submitted 2015-01-06; First posted 2015-01-15 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2017-08

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ventilation during labor analgesia: We are simply measuring ventilation changes that occur following labor analgesia.
  Interventions: Other: Labor analgesia

INTERVENTIONS:
Other: Labor analgesia — Measuring maternal ventilation after placement of epidural analgesia compared to baseline

SUMMARY:
Epidural techniques offer the advantage of being able to titrate the level, density, and duration of the blockade through the use of a catheter and are associated with relative maternal hemodynamic stability. One of the disadvantages, however, include a raise in maternal temperature that is attributed to labor epidural technique. This study will assess if decreased maternal ventilation following induction of labor analgesia causes a raise in temperature.

DETAILED DESCRIPTION:
Fever in labor complicates up to one-third of deliveries. The etiologies of intrapartum fever are diverse and include maternal chorioamnionitis, and other infections. In addition, epidural analgesia used for pain relief in labor is associated with mild maternal temperature increase and overt fever. Originally dismissed by obstetric anesthesiologists as a clinical curiosity of little consequence, epidural-associated hyperthermia may lead to significant maternal as well as fetal or neonatal adverse effects. Observational investigations performed 2 decades ago demonstrated a gradual increase in temperature in laboring parturients with epidural analgesia not see in those electing systemic opioid analgesia or no analgesia. The epidural group showed an average increase in temperature of approximately 1 degree centigrade over 7 hours whereas temperatures in non-epidural group remained constant. No evidence of clinical infection was reported in any of the women. Many studies confirmed these raises in temperature in epidural group compared to no epidural group during labor and delivery.

Several mechanisms have been postulated with no study reaching a conclusion. The mechanisms suggested include imbalance between heat production and heat dissipation, effect of opioid on interleukin-2, markers of inflammation induced by epidural analgesia, etc. Our study aims at the first mechanism. It may be a physiological process that leads to an imbalance between heat production and heat dissipation. Labor is a hyper metabolic state and increased heat production is dissipated via increased ventilation that is associated with labor pains with no epidural pain relief. It is conceivable that laboring women with pain relief subsequent to epidural analgesia, a decrease in ventilations may occur leading to decreased heat dissipation.

ELIGIBILITY:
Inclusion Criteria:

1. Parturient with no major co-morbidities
2. Singleton, vertex gestation at term (38-42 weeks)
3. Less than 5 cm dilation
4. Intact fetal membranes or rupture for < 6 hrs.
5. Desire to have an epidural technique for labor analgesia

Exclusion Criteria:

1. Current or historical evidence of clinically significant disease or condition, including diseases of pregnancy (i.e preeclampsia, gestational diabetes)
2. Any contraindication to the administration of an epidural technique
3. History of hypersensitivity or idiosyncratic reaction to local anesthetic or opioid medications
4. Current or historical evidence of a disease which may result in the risk of a cesarean delivery (i.e. vaginal birth after cesarean section, history of uterine rupture)
5. Evidence of anticipated fetal anomalies
6. Signs or symptoms consistent with an infection or sepsis; baseline temperature < 37 degrees Celsius, or 99 degrees Fahrenheit.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Informed consent will be obtained by one of the licensed physician investigators at the earliest opportunity when the subject arrives on the labor suite and following contact with their provider. While the timing between subject arrival and request for neuraxial analgesia can be variable, in subjects who present in early labor at less than 5 cm cervial dilation, there is often several hours available for a subject to consider 1) whether they desire a central neuraxial technique during labor, and 2) whether they would be willing to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2014-08-14 (Actual); Primary Completion 2016-09-02 (Actual); Study Completion 2016-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhavani Kodali, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kodali BS, Choi L, Chau A, Harvey BC, Brayanov J, Tsen LC, Palanisamy A. Use of a novel non-invasive respiratory monitor to study changes in pulmonary ventilation during labor epidural analgesia. J Clin Monit Comput. 2020 Jun;34(3):567-574. doi: 10.1007/s10877-019-00349-1. Epub 2019 Jul 8. PMID 31286333

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following approval by our Institutional Review Board, written consent was obtained from 57 healthy, full-term women undergoing elective induction of labor who expressed interest in receiving epidural analgesia.
Groups:
- Study Group: Maternal ventilation was measured non-invasively using the ExSpiron Respiratory Volume Monitor (RVM) in forty-one term parturients who received labor epidural analgesia. Minute ventilation (MV), respiratory rate (RR), and tidal volume (TV) were measured via chest pads using bio-impedance technology. In addition, we recorded vital signs and maternal oral temperature at 5, 10, 15, 20, 25, 30 and 60 min after epidural analgesia initiation, and then every hour until delivery.
Period: Overall Study
Arm/Group | Study Group
Started | 57
Completed | 41
Not Completed | 16

BASELINE CHARACTERISTICS:
Groups:
- Study Group: We are simply measuring ventilation changes that occur following labor analgesia.
  Labor analgesia: Measuring maternal ventilation after placement of epidural analgesia compared to baseline
Arm/Group | Study Group
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 57
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Changes in Maternal Ventilation During Labor Analgesia
Description: If Maternal Ventilation decreases following labor analgesia at 2 hour and 4 interval
Time Frame: Ventilation parameters measured at 2 hour and 4 hour
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Study Group
Number analyzed (Participants) | 41
L/min
  Maternal ventilation at baseline | 15.3 (1)
  Maternal ventilation at 2 hours | 12.6 (1.1)
  Maternal Ventilation at 4 hor | 13.8 (1.2)

2. Secondary Outcome: If Maternal Temperature Increases During Labor Analgesia
Description: If maternal temperature increases during labor analgesia
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: Degree F
Arm/Group | Ventilation During Labor Analgesia
Number analyzed (Participants) | 41
Degree F
  baseline temperature | 98.1 (0.4)
  Temperature at 4 hour | 98.7 (0.5)

ADVERSE EVENTS:
Time Frame: Only for the study period
Description: No adverse events observed
Arm/Group | Ventilation During Labor Analgesia
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No